CLINICAL TRIAL: NCT06793462
Title: ASSESSMENT of FRAILTY AS a PROGNOSTIC FACTOR for MORTALITY, DISABILITY, and QUALITY of LIFE AFTER ICU ADMISSION
Acronym: FG-UCI
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)348/2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Frailty At Older Adults
Keywords: FRAILTY AND ICU; PROGNOSTIC; ELDERLY; FUNCTIONAL; QUALITY OF LIFE
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FRAILS AND NO FRAILS

SUMMARY:
Between 30% and 40% of elderly patients (over 70 years old) who require hospitalization and treatment in Intensive Care Units (ICU) exhibit a state of frailty. This condition is associated with adverse prognostic factors such as increased in-hospital mortality, functional decline, and a deterioration in their long-term quality of life. Some frail elderly patients may require invasive mechanical ventilation (ventilator) as life support during the acute phase, which has also been linked to adverse prognostic outcomes. Additionally, frailty is common in patients with severe infections, with a high mortality rate, subsequent functional decline, and reduced quality of life following ICU admission.

DETAILED DESCRIPTION:
This project focuses on evaluating the role of geriatric frailty (FG) as a crucial predictive factor in various clinical aspects of elderly patients requiring admission to intensive care units (ICUs). Below is a breakdown of the project's main objectives for clarity:

Frailty as a predictor of mortality:

Assess whether frailty is an independent marker that predicts mortality over different timeframes (short, medium, and long term) in elderly patients admitted to the ICU.

Frailty and functional disability:

Determine whether frailty is associated with the evolution of functional disability in the short, medium, and long term following ICU admission.

Frailty and quality of life:

Analyze whether frailty can predict changes in the quality of life of elderly patients after their stay in the ICU, considering the same timeframes (short, medium, and long term).

Impact on patients requiring invasive mechanical ventilation (IMV):

Evaluate the impact of frailty on mortality, functional evolution, and quality of life in elderly patients requiring IMV.

Study the role of frailty as a prognostic factor for complications related to weaning from mechanical ventilation (tracheostomy, prolonged ICU or hospital stay, readmissions, and disability).

Frailty and sepsis/septic shock:

Investigate whether frailty is an independent prognostic marker for mortality in elderly patients with sepsis or septic shock admitted to the ICU.

This comprehensive approach aims not only to identify frailty as a key risk factor but also to guide management strategies and clinical decision-making for this particularly vulnerable population. If you need further elaboration or scientific drafting, feel free to ask!

ELIGIBILITY:
Inclusion criteria:

* Elderly patients over 70 years of age requiring admission to ICU-semicritical units.
* Patients receiving at least one life-support intervention for more than 24 hours, including:
* Mechanical ventilation (invasive or non-invasive),
* Vasopressor or inotropic treatment,
* Requirement for acute renal replacement therapies for more than 24 hours,

Extracorporeal support such as:

Veno-Venous Extracorporeal Membrane Oxygenation (ECMO-VV), Veno-Arterial Extracorporeal Membrane Oxygenation (ECMO-VA).

Exclusion Criteria:

* Patients with an ICU stay of less than 72 hours.
* Patients with treatment limitations upon ICU admission, although an isolated "Do Not Resuscitate" (DNR) order is acceptable; life expectancy of less than 6 months.
* Absence of family members or caregivers available to provide medical history. Language barriers (non-Spanish speakers without access to medical translators).
* Structural neurological diseases requiring ICU admission, including stroke or spinal cord pathology.
* Patients for whom 12-month follow-up is anticipated to be unfeasible.
* Patients without consent authorization.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population will consist of all elderly patients (over 70 years old) requiring admission to ICU-Semi-critical units, with consecutive sampling for the treatment of life-threatening conditions based on the following selection criteria:
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
MORTALITY | ONE YEAR
  Determine whether frailty is a predictor of short-, medium-, and long-term mortality in elderly patients requiring ICU admission.